CLINICAL TRIAL: NCT02509481
Title: Repeat Ivermectin Mass Drug Administrations for Control of Malaria: a Pilot Safety and Efficacy Study
Acronym: RIMDAMAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); Centre Muraz (Other); Ministère de la Santé du Burkina Faso (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5375011; OPP1116536 (Other Grant/Funding Number: The Bill and Melinda Gates Foundation)
Record Dates: First submitted 2015-07-23; First posted 2015-07-28 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Malaria; Lymphatic Filariasis
Keywords: malaria; lymphatic filariasis; mosquito; ivermectin; mass drug administration
MeSH Terms: conditions — Malaria; Elephantiasis, Filarial | interventions — Ivermectin; Albendazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single MDA (Active Comparator): Single mass drug administration of ivermectin (150 µg/kg) + albendazole (400 mg) performed after the start of the rainy season as part of public health efforts to eliminate lymphatic filariasis.
  Interventions: Drug: Ivermectin; Drug: Albendazole
- Repeated MDA (Experimental): Same at Active Comparator, but then followed by five more mass drug administrations of ivermectin only (150 µg/kg) every three weeks thereafter.
  Interventions: Drug: Ivermectin; Drug: Albendazole

INTERVENTIONS:
Drug: Ivermectin
  Other Names: Mectizan
Drug: Albendazole

SUMMARY:
The purpose of this study is to determine whether repeated ivermectin mass drug administrations to Burkinabé villagers, performed in three week intervals over the rainy-season, is well-tolerated and safe, and also effective in reducing local malaria transmission and thus clinical malaria episodes in treated village children.

DETAILED DESCRIPTION:
Primary Objective: To determine the efficacy of repeated ivermectin mass drug administrations (IVM MDA) (150 µg/kg), given to the population of eligible patients in enrolled villages, for reducing the cumulative incidence of uncomplicated malaria episodes in enrolled village children (≤ 5 years of age) over the course of the treatment.

Hypothesis: Repeated IVM MDA starting at the beginning of the rainy season will be well tolerated and safe, and will reduce clinical malaria episodes in children by significantly reducing malaria transmission among treated villages.

Overview Study Design: Single-blind (outcomes assessor); parallel assignment with 2 arms; cluster-randomized control trial to determine the effect of repeated IVM MDA on malaria transmission and clinical malaria episodes. The unit of randomization will be the village (cluster). 8 villages total will be enrolled in two arms. The active comparator arm (4 villages) will receive a single standard MDA (IVM; 150-200 µg/kg + albendazole; 400 mg) soon after the start of the rainy season, while the experimental arm (4 villages) will receive the standard MDA on the same date, plus 5 more IVM MDA at 3 week intervals thereafter. The primary endpoint will be the cumulative incidence of clinical malaria episodes in children ≤5 year of age within each village.

Sites: This study will be conducted in villages along the main east-west and north-south road corridors in the Sud-Ouest administrative region of Burkina Faso.

Study Population: Indigenous Burkinabé from various ethnic groups (Dagara, Bobo, Lobi, Mossi, etc.). The entire eligible population of each enrolled village will receive the MDAs, following the standard inclusion/exclusion criteria of MDA for control of microfilaremia caused by Wuchereria bancrofti (lymphatic filariasis; LF). Clinical incidence of malaria will be assessed only in children living in enrolled villages who are ≤ 5 years of age, most of whom will not have received any treatment due to the standard MDA exclusion criteria of children < 90 cm.

Study Interventions: 2 arms: 1) Active comparator arm - single standard MDA with IVM (150 µg/kg) + albendazole (ALB;400 mg) soon after the beginning of the rainy season; 2) Experimental arm, single standard MDA with IVM (150 µg/kg) + ALB (400 mg) plus 5 more MDA with IVM alone (150 µg/kg) at 3 week intervals thereafter. Community health workers and trained by local health authority of the Sud-Ouest region will perform the first MDA in both arms with logistical assistance from the study investigators. Repeated MDAs will only occur in the experimental-arm villages, and be performed by the study investigators.

Follow-up Procedures: Trained nurses will visit each study village each week over the course of the study to investigate and record any adverse events or severe adverse events communicated by the study population. They will also perform active case surveillance each week on enrolled village children for clinical malaria episodes, defined as ≥38.0°C fever or history of fever in the last 24 hours + positive rapid diagnostic test for Plasmodium falciparum. Secondary measures will be collected by the nurses.

Sample Size: Assuming an 80% cumulative incidence of malaria episodes in the control arm and an intracluster correlation coefficient of 0.02, 4 clusters are needed per arm and 69 children enrolled per cluster to detect a conservative 40% reduction in incidence in the treatment arm with 80% power and a statistical confidence of 95%.

Safety Outcomes:

• Adverse events (seriousness, causality, expectedness)

Secondary Outcomes:

* Incidence of new P. falciparum infections acquired (molecular force-of-infection)
* Prevalence and intensity (eggs/larvae per gram of feces) of soil transmitted helminth infections in a subset of treated patients between 6-10 years of age.
* Indoor-resting Anopheles mosquito capture rate
* Outdoor-host seeking Anopheles mosquito capture rate
* Adult mosquito age structure (parity rate) in captured mosquitoes
* Plasmodium sporozoite rate/entomological inoculation rate in captured mosquitoes
* Rate of Wuchereria bancrofti in captured mosquitoes

ELIGIBILITY:
Inclusion Criteria:

* Residence in the study site
* Able to understand the information and willing to give consent and assent (parent or guardian consent if study participant age is < 18 years)

Exclusion Criteria:

* Residence outside of in the study site
* Height ≤ 90 cm
* Permanent disability, serious medical illness that prevents or impedes study participation and/or comprehension
* Pregnancy
* Breast feeding if infant is within 1 week of birth
* Known allergy to the study drugs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2712 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian D. Foy, PhD, Principal Investigator — Colorado State University; Roch K Dabire, PhD, Principal Investigator — Institute de Recherche en Sciences de la Santé
Locations (2):
- Colorado State University, Fort Collins, Colorado, United States
- Institut de Recherche en Sciences de la Santé, Bobo-Dioulasso, Houet, Burkina Faso

REFERENCES:
- [Derived] Foy BD, Alout H, Seaman JA, Rao S, Magalhaes T, Wade M, Parikh S, Soma DD, Sagna AB, Fournet F, Slater HC, Bougma R, Drabo F, Diabate A, Coulidiaty AGV, Rouamba N, Dabire RK. Efficacy and risk of harms of repeat ivermectin mass drug administrations for control of malaria (RIMDAMAL): a cluster-randomised trial. Lancet. 2019 Apr 13;393(10180):1517-1526. doi: 10.1016/S0140-6736(18)32321-3. Epub 2019 Mar 14. PMID 30878222

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2712 participants from 8 villages were recruited to participate and enrolled. Importantly, the intervention (repeated ivermectin MDA) was given to most villagers and the safety outcome was assessed in this whole group. However, the primary outcome was assessed in a cohort of 590 enrolled village children ≤5 years old.
Groups:
- Single MDA: Single mass drug administration of ivermectin (150 µg/kg) + albendazole (400 mg) performed after the start of the rainy season as part of public health efforts to eliminate lymphatic filariasis.
  Ivermectin
  Albendazole
- Repeated MDA: Same as Active Comparator, but then followed by five more mass drug administrations of ivermectin only (150 µg/kg) every three weeks thereafter.
  Ivermectin
  Albendazole
Period: Overall Study
Arm/Group | Single MDA | Repeated MDA
Started | 1265 | 1447
Completed | 1265 | 1447
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The total number of enrolled participants were most of population of the eight enrolled villages (2712 participants).
Groups:
- Total: Total of all reporting groups
Arm/Group | Single MDA | Repeated MDA | Total
Number analyzed (Participants) | 1265 | 1447 | 2712
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14 [7 to 30] | 16 [6 to 35] | 15 [6 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 620 | 713 | 1333
  Male | 645 | 734 | 1379
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1265 | 1447 | 2712
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Burkina Faso | 1265 | 1447 | 2712
Height <90 cm [Count of Participants; unit: Participants] | 210 | 267 | 477

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Clinical Malaria Episodes
Description: Cumulative incidence of malaria episodes in a cohort of village children ≤ 5 years of age (as assessed by active case surveillance in study villages - malaria episode defined as ≥38.0°C fever or history of fever in the last 24 hours + positive rapid diagnostic test for Plasmodium falciparum). Incidence is reported as malaria episodes per child over the course of the trial, a higher incidence is a worse outcome.
Time Frame: Approximately 18 weeks, from the start of the first MDA to 3 weeks following the last MDA in the Experimental arm
Population: Note that the primary outcome measure comes only from malaria incidence measurements within this child cohort (590 children). It is not a measure of malaria incidence from all enrolled participants from the study villages (2712 participants).
Measure: Mean (95% Confidence Interval); unit: episodes
Arm/Group | Single MDA | Repeated MDA
Number analyzed (Participants) | 263 | 327
episodes | 2.49 [2.28 to 2.73] | 2.00 [1.82 to 2.20]

2. Secondary Outcome: Adverse Events
Description: The number of adverse events. Adverse events data were collected via passive case detection from total population.
Time Frame: Approximately 18 weeks, from the start of the first MDA to 3 weeks following the last MDA in the Experimental arm
Population: Per protocol, the secondary outcome was a measure of all adverse events, excluding uncomplicated malaria episodes that were reported in the primary outcome, that occurred among the total enrolled population from the study villages (2712 participants).
Measure: Number; unit: adverse events
Arm/Group | Single MDA | Repeated MDA
Number analyzed (Participants) | 1265 | 1447
adverse events | 24 | 45

3. Secondary Outcome: Entomological Indicator of Parasite Transmission
Description: Change in human IgG reactivity (optical density; ∆OD) to an Anopheles salivary gland antigen (peptide gSG6-P1) over the trial period. A score of 0 indicates no change in seroreactivity from from immediately before to immediately after the trial, suggesting consistent mosquito biting throughout the trial. A positive score indicates increasing seroreactivity and thus increasing mosquito biting on participants from immediately before to immediately after the trial. A negative score indicates decreasing seroreactivity and thus decreasing mosquito biting on participants from immediately before to immediately after the trial.
Time Frame: Approximately 20 weeks, from before the start of the first MDA to 4 weeks following the last MDA in the Experimental arm
Population: We sampled finger capillary blood pre-intervention from a subset of enrolled participants located in 8 households at the center of each study village, and then re-sampled their blood immediately after the intervention period. Data were reported only from participants that gave both sets of samples (221 of 2712 participants).
Measure: Mean (95% Confidence Interval); unit: change in IgG ELISA optical density
Arm/Group | Single MDA | Repeated MDA
Number analyzed (Participants) | 95 | 126
change in IgG ELISA optical density | -0.057 [-0.096 to -0.017] | -0.124 [-0.161 to -0.088]

4. Secondary Outcome: Molecular Force of P. Falciparum Infection
Description: Examination of new P. falciparum clones acquired from the beginning to the end of the intervention (molecular force of infection; mFOI) per child. Molecular genotyping used capillary blood taken at the time of diagnosis of each positive malaria episode and consisted of nPCR of the msp2 gene. We calculated the multiplicity of infection (MOI) per malaria episode, and then calculated the molecular force of infection (mFOI) associated with malaria episodes per child (over course of the trial)
Time Frame: Approximately 18 weeks, from the start of the first MDA to 3 weeks following the last MDA in the Experimental arm
Population: Molecular genotyping was performed on blood samples from 132 enrolled cohort children who were selected using a random sequence generator. Genotyping was successful on blood spots corresponding to 153 malaria episodes, which allowed us to calculate the mFOI over the trial from 76 enrolled children from the cohort.
Measure: Median (Inter-Quartile Range); unit: new P. faliciparum infections per child
Arm/Group | Single MDA | Repeated MDA
Number analyzed (Participants) | 38 | 38
new P. faliciparum infections per child | 4 [2 to 7] | 3 [2 to 5]

5. Secondary Outcome: Number of 6-10 Year Old Participants With Soil Transmitted Helminths (STH)
Description: Prevalence of soil transmitted helminth infections in children between 6-10 years old from the beginning to the end of the intervention
Time Frame: as for outcome 3
Population: This outcome was only measured in older enrolled children between 6-10 years of age, who were not in our primary outcome cohort, and who were eligible to be treated with ivermectin due to their height >90 cm (232 of 2712 participants).
Measure: Number; unit: participants
Arm/Group | Single MDA | Repeated MDA
Number analyzed (Participants) | 122 | 110
participants | 3 | 0

6. Secondary Outcome: Entomological Inoculation Rate
Description: The entomological inoculation rate (EIR per week per person) is the measure of the human biting rate per person per week, multiplied by the sporozoite rate (in biting mosquitoes) per week, an estimated from sampling mosquitoes from 8 households located in the center of each study village. The EIR was calculated for each of the 6 sampling weeks of the treatment phase.
Time Frame: 6 sampling periods over 18 weeks, starting in week 2 following the first MDA, and sampling every 3 weeks thereafter until week 17 of the treatment phase.
Population: The mean EIR was calculated across the 6 sampling periods in the 8 study villages (4 villages in each arm). EIR was calculated from the number of mosquitoes captured in select houses and the number of enrolled participants who lived in each sampled house (324/1265 in single MDA arm, and 271/1447 in repeated MDA arm).
Measure: Mean (Standard Deviation); unit: infectious bites per person per week
Arm/Group | Single MDA | Repeated MDA
Number analyzed (Participants) | 324 | 271
infectious bites per person per week | 0.2069 (0.2376) | 0.1972 (0.2084)

ADVERSE EVENTS:
Description: Adverse events were measured from the total population of enrolled participants in the eight study villages (n=2712), and most of these participants received the study intervention (ivermectin MDA)
Arm/Group | Single MDA | Repeated MDA
All-Cause Mortality (participants affected / at risk) | 5/1265 | 15/1447
Serious Adverse Events (participants affected / at risk) | 10/1265 | 19/1447
Other Adverse Events (participants affected / at risk) | 14/1265 | 26/1447
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single MDA (N=1265) | Repeated MDA (N=1447)
moderate to severe malaria (Infections and infestations) | 7 (7) | 7 (7)
neonatal infection (Infections and infestations) | 1 (1) | 0 (0)
untreated decompensated hypertensive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
fever, vomiting, anorexia (Infections and infestations) | 1 (1) | 0 (0)
acute intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
liver disease: ascites + bulky edema of the lower limbs. (Hepatobiliary disorders) | 0 (0) | 1 (1)
liver cancer, cirrhosis of the liver (Hepatobiliary disorders) | 0 (0) | 1 (1)
abdominal pain, loose stool, vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
fever, anemia, cachexia (Infections and infestations) | 0 (0) | 1 (1)
severe sepsis (Infections and infestations) | 0 (0) | 1 (1)
unspecified sudden death in the early morning (Investigations) | 0 (0) | 1 (1)
vomiting, hematemesis, bloody stool, cardiovascular shock (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal bloating, fecal matter obstruction, anuria, refusal to breastfeed (Gastrointestinal disorders) | 0 (0) | 1 (1)
fever and chills; suspected typhoid fever (Infections and infestations) | 0 (0) | 1 (1)
snakebite envenomation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infectious pneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single MDA (N=1265) | Repeated MDA (N=1447)
malaria (Infections and infestations) | 2 (2) | 2 (2)
acute malnutrition (Infections and infestations) | 2 (2) | 5 (5)
fever (Infections and infestations) | 1 (1) | 0 (0)
diarrhea (Infections and infestations) | 1 (1) | 0 (0)
unspecified injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
stage 3 tooth decay with local tumefaction (Infections and infestations) | 1 (1) | 0 (0)
Bilateral palpebral edema (Eye disorders) | 1 (1) | 0 (0)
Tremor, palpitations, arthralgia (General disorders) | 1 (1) | 0 (0)
Perforated bilaterally suppurated otitis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
pruritis (Immune system disorders) | 1 (1) | 2 (2)
snakebite envenomation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
intercostal zoster from immune system depression (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
acute otitis media (Ear and labyrinth disorders) | 0 (0) | 1 (1)
febrile diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
first degree burn over 80% of lower right limb (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
suppurative otitis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
unspecified injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Involuntary abortion at two months of pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
road accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chronic wound in the left ankle (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
(General disorders) | 0 (0) | 1 (1)
Postpartum pelvic pain (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abdominal pain, loose stool, vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
headache and chills; suspected infectious origin (Infections and infestations) | 0 (0) | 1 (1)
Swelling of the feet, hyperthermia and chills (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
fever and chills; suspected typhoid (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
We could not provide placebo MDA for the control villages, and the trial was not blinded to the study population or the study team. Adverse event analysis bias may have from the knowledge of the village populace as to what arm they were part of.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-07-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT02509481/Prot_SAP_ICF_000.pdf